CLINICAL TRIAL: NCT00004577
Title: Characterization of Brain Morphology and Activity Using Functional and Anatomical MRI Contrast
Brief Title: Study of New Magnetic Resonance Imaging Methods of the Brain
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000082; 00-N-0082
Record Dates: First submitted 2000-02-18; First posted 2000-02-21 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01-12

CONDITIONS: Healthy Volunteer; Magnetic Resonance Imaging; Healthy; fMRI; Brain Mapping; Adult
Keywords: Brain Morphology; Cerebral Blood Volume; Functional Imaging; Development; MEG; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteer: Any healthy, male or female volunteer 18 years of age and older.

SUMMARY:
The purpose of this investigation is to develop improved magnetic resonance imaging (MRI) techniques and hardware for studying brain function. MRI is a diagnostic tool that provides information about brain chemistry and physiology. This study will evaluate new MRI methods for monitoring blood flow to regions of the brain in response to simple tasks. The MRI machine used in this study is more powerful than those in most hospitals, permitting a higher visual resolution.

Normal healthy volunteers over 18 years old may be eligible for this study. Candidates will be screened with a medical history and questionnaire, and a neurological examination. Study participants will have a yearly MRI scan. For this procedure, the subject lies on a stretcher that is moved into a donut-shaped machine with a strong magnetic field. A lightweight circular or rectangular coil a device that improves the quality of the images may be placed on the head. The scan time varies from 20 minutes to 3 hours; most scans last between 45 and 90 minutes. During the scan, the subject may perform simple tasks, such as listening to tapes, tapping a finger, moving a hand, watching a screen, or smelling a fragrance. More complex tasks may require thinking about tones or pictures and responding to them by pressing buttons.

Information from this study will be used to develop better imaging methods that will, in turn, permit a greater understanding of normal and abnormal brain behaviors.

DETAILED DESCRIPTION:
Objective

The goal of this protocol is to improve spatial resolution and contrast in MRI studies of brain anatomy and function, by developing novel hardware, and image acquisition and reconstruction techniques. Specifically, by improving MRI image quality and manipulating MRI contrast, we aim to better characterize and quantify structural, chemical, and blood flow variations across the brain, and study their relationship with neuronal activity. For this purpose, we will develop and optimize novel MRI techniques on normal, healthy volunteers, and combine these with EEG and recording of other physiological signals.

Study Population

Any healthy, male or female volunteer 18 years of age and older; the subjects must be capable of understanding the procedures and requirements of this study and be willing to sign an informed consent document.

Design

This is a technical development study design to develop and evaluate new MR technology for performing MRI and functional MRI in the CNS with novel contrasts and with a high spatial resolution.

Outcome Measures

The primary outcome of this study will be the ability to acquire anatomical and functional images of the human brain with high spatial resolution, i.e., 200-500 micron and 750-1000 micron respectively. In addition, developed techniques will allow the robust measurement of specific tissue properties, including diffusion, structural anisotropy, iron and myelin content, perfusion, and metabolite concentrations. The relative merits of blood flow and blood oxygenation level dependent (BOLD) functional MRI (fMRI) techniques, and their particular spatial and temporal signal characteristics will be established. It will be determined whether information valuable to interpret BOLD fMRI can be derived from EEG and other physiological signals.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18 years of age and older
* in good general health
* able to understand the procedures and requirements and give informed consent

EXCLUSION CRITERIA:

All Subjects will undergo a neurological physical and answer the Healthy volunteer form, and the most-recent version of the NMR safety screening form

A subject will be excluded if he/she:

1. has any metal implant or objects of unknown identity or composition, or if it s known to be non-compatible with MRI, such as pacemakers, medication pumps, aneurysm clips, metallic prosthesis (such as heart valves or cochlear implants), certain orthopedic implants (pins and rods), shrapnel, or small metal fragments in the eye;
2. has claustrophobia;
3. cannot lie comfortably for up to 120 minutes;
4. underwent brain surgery or suffered a traumatic head trauma;
5. has migraines that require medication;
6. has ever been hospitalized for a psychiatric disorder;
7. has medical health problems such as pulmonary or airway disease, heart failure, coronary artery disease, and uncontrolled hypertension which would require physiological monitoring during the scan;
8. has a history of any medical condition that could result in an emergency medical situation while undergoing the MRI scan;
9. has hearing problems which would make it difficult to tolerate scanner noise;
10. is pregnant;
11. has body/make-up tattoos (e.g. lips, eyebrows, eyeliner). Each tattoo will be considered on a case-to-case basis, taking into account of the age and location of the tattoo;
12. has a sleep apnea diagnosis;
13. has a neurological disorder, such as Stroke, Parkinson s, and Epilepsy;
14. a member of the NINDS Laboratory of Functional and Molecular Imaging.

The contraindications to MRI at the various field strengths are almost identical, except the 7 T also excludes subjects with gold dental crowns.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteer
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2000-07-01 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to develop and evaluate new MR pulse sequences and hardware for performing anatomical and functional MRI in the CNS at, 3.0T, and 7T with a high spatial resolution. | annually
  The primary outcome of this study will be the ability to robustly acquire whole brain MRI sensitized to myelin, iron, diffusion, perfusion, and fiber orientation. Perfusion- and BOLD- based fMRI techniques will allow distinguishing between neuronal and systemic vascular signal contributions. In addition, we anticipate the ability to acquire (proton) spectroscopic data at 5mm resolution.

SECONDARY OUTCOMES:
To develop an understanding of the limits in contrast and resolution of anatomical and functional MRI.To develop an understanding of the merits of high field MRI for the study of brain anatomy and function. | annually
  Secondary outcome measure will be an estimate of the relative performance levels of the different field strengths for anatomical, functional and spectroscopic imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Alan P Koretsky, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogawa S, Lee TM, Kay AR, Tank DW. Brain magnetic resonance imaging with contrast dependent on blood oxygenation. Proc Natl Acad Sci U S A. 1990 Dec;87(24):9868-72. doi: 10.1073/pnas.87.24.9868. PMID 2124706
- [Background] Ogawa S, Tank DW, Menon R, Ellermann JM, Kim SG, Merkle H, Ugurbil K. Intrinsic signal changes accompanying sensory stimulation: functional brain mapping with magnetic resonance imaging. Proc Natl Acad Sci U S A. 1992 Jul 1;89(13):5951-5. doi: 10.1073/pnas.89.13.5951. PMID 1631079
- [Background] Detre JA, Leigh JS, Williams DS, Koretsky AP. Perfusion imaging. Magn Reson Med. 1992 Jan;23(1):37-45. doi: 10.1002/mrm.1910230106. PMID 1734182
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-N-0082.html